CLINICAL TRIAL: NCT00001382
Title: A Phase I Study of Recombinant Vaccinia Virus That Expresses Prostate Specific Antigen in Adult Patients With Adenocarcinoma of the Prostate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940118; 94-C-0118
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Prostatic Neoplasms
Keywords: Immunotherapy; Vaccine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC

INTERVENTIONS:
Biological: PROSTVAC

SUMMARY:
This trial will evaluate, in patients with metastatic prostate cancer, the tolerability, toxicities, efficacy, and immunologic effects of repeated vaccinations with a recombinant vaccinia virus that contains the Prostate Specific Antigen gene (PROSTVAC).

DETAILED DESCRIPTION:
This trial will evaluate, in patients with metastatic prostate cancer, the tolerability, toxicities, efficacy, and immunologic effects of repeated vaccinations with a recombinant vaccinia virus that contains the Prostate Specific Antigen gene (PROSTVAC). Patients with PSA-expressing adenocarcinoma of the prostate will be evaluated for eligibility that includes a history of prior vaccinia (as vaccine against smallpox) and immunocompetence. We completed a phase I trial investigating the use of rV-CEA in adenocarcinomas of the GI tract, lung and breast. The toxicities encountered are local reactions to the vaccine. We did not encounter any myelosuppression or systemic autoimmune reaction. We would like to evaluate four doses to ensure safety and to decide a best biological dose. Six patients will receive 2.65 x 10(5) PFU and 2.65 x 10(6) PFU of vaccine by scarification. Because higher doses cannot be achieved by scarification, six patients will receive 2.65 x 10(7) PFU and 2.65 x 10(8) PFU subcutaneously. We plan to give three vaccinations at four week intervals. All six patients treated in each dose level must be evaluable for 4 weeks before enrolling patients at the higher dose level. No intrapatient escalation is planned. Toxicity, tumor response, and humoral and cellular immunity factors will be monitored. Optional lymphapheresis will be done on patients that are HLA A2. Once we determined the best biological dose, we would like to accrue an additional 6 patients to that level.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically confirmed adenocarcinoma of the prostate as follows: Unresectable and/or incurable tumor AND Tumor progression after at least 1 prior hormonal manipulation (i.e., LHRH agonist/flutamide or orchiectomy). LHRH agonist may by continued concurrently with protocol therapy.

New bone or soft tissue lesions OR Serum PSA that has risen on 3 successive evaluations at least 1 week apart during and/or after hormonal therapy. If PSA is below 4 ng/mL, measurable disease with positive immunohistochemical stain for PSA is required.

No history of allergy to eggs.

No history of or active CNS metastases.

Symptomatic spinal or other bony metastasis should be irradiated prior to entry.

Bi-dimensionally measurable disease not required.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy:

No concurrent Biologic Therapy.

Must fully recover from prior Biologic Therapy.

Chemotherapy:

At least 4 weeks since prior chemotherapy and fully recovered.

No more than 1 prior chemotherapy regimen.

No concurrent chemotherapy.

Endocrine Therapy:

See Disease Characteristics.

At least 4 weeks since prior hormonal therapy and fully recovered.

No concurrent steroids.

Radiotherapy:

At least 4 weeks since prior radiation therapy and fully recovered.

No prior radiotherapy to more than 50% of nodal groups.

No concurrent radiotherapy.

Surgery:

At least 4 weeks since prior surgery, with surgical scar healed.

No prior splenectomy.

PATIENT CHARACTERISTICS:

Age: Over 18.

Performance status: Zubrod (ECOG) 0-2.

Hematopoietic:

Absolute granulocyte count greater than 2,000/mm(3);

Platelet count greater than 100,000/mm(3);

Hemoglobin greater than 8.0 g/dL.

Hepatic:

Bilirubin less than 1.6 mg/dL;

AST and ALT less than 4 times normal.

Renal: Creatinine less than 1.6 mg/dL.

Immunologic:

Prior vaccinia (for smallpox immunization) required, with proof of vaccination as follows: Detectable anti-vaccinia antibodies, Physician certification of prior vaccination, Patient recollection or appropriate vaccination-site scar sufficient in patients over age 25, Delayed-type hypersensitivity skin testing (to mumps, Candida, and Trichophyton antigens) normal Quantitative immunoglobulins normal.

No evidence of immunocompromise, i.e.:

No HIV antibody;

No eczema or atopic dermatitis;

No autoimmune neutropenia, thrombocytopenia, or hemolytic anemia;

No systemic lupus erythematosus, Sjogren syndrome, or scleroderma;

No myasthenia gravis;

No Goodpasture syndrome;

No Addison's disease, Hashimoto's thyroiditis, or active Graves' disease;

No other autoimmune disease or diagnosis of altered immune function.

OTHER:

No active case or history of extensive psoriasis, severe acneiform rash, impetigo, varicella zoster, burns, or other traumatic or pruritic skin condition.

No active infection requiring antibiotics (including chronic suppressive therapy). At least 3 days since antibiotic therapy.

No history of seizures, encephalitis, or multiple sclerosis.

No other serious intercurrent illness.

Able to avoid close contact with the following individuals for at least 2 weeks after vaccination (i.e., no such individuals as household members and no care-giving responsibilities for such individuals): Children under age 3, Pregnant women, Individuals with eczema or skin conditions defined above, Leukemia or lymphoma patients, HIV-positive individuals, Patients receiving immunosuppressive therapy, Any other immunosuppressed individuals.

No prior malignancy unless curatively treated and patient has been in remission for at least 2 years (excluding squamous cell or basal cell carcinoma of the skin or carcinoma in situ of the cervix).

Able and willing to travel to the NIH, NCI-NMOB, or the Lombardi Cancer Center at Georgetown University for treatment and follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1994-03; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States